CLINICAL TRIAL: NCT05194982
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-B01D1 in Patients With Locally Advanced or Metastatic Solid Tumor
Brief Title: A Study of BL-B01D1 in Patients With Locally Advanced or Metastatic Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-101
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Solid Tumor
Keywords: Non-Small Cell Lung Cancer (NSCLC); Small cell lung cancer (SCLC); Nasopharyngeal cacinoma (NPC); Head and Neck Cancer (HNC)
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
In phase Ia study, the safety and tolerability of BL-B01D1 in patients with locally advanced or metastatic solid tumor will be investigated to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) of BL-B01D1.

In phase Ib study, the safety and tolerability of BL-B01D1 at the phase Ia recommended dose will be further investigated, and recommended phase II dose (RP2D) for phase II clinical studies will be determined.

In addition, the preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of BL-B01D1 in patients with locally advanced or metastatic solid tumor will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign the informed consent form voluntarily and follow the plan requirements.
2. No gender limit.
3. Age: ≥18 years old and ≤75 years old (stage Ia); ≥18 years old (stage Ib).
4. Expected survival time ≥ 3 months.
5. Locally advanced or metastatic solid tumor confirmed by histopathology and/or cytology, which are incurable or currently without standard treatment.
6. Agrees to provide archived tumor tissue specimens or fresh tissue samples from the primary lesion or metastasis within 2 years; If a subject is unable to provide a tumor tissue sample, he/she may be enrolled after being evaluated by the investigator if other inclusion criteria are met.
7. Participants must have at least one measurable lesion that meets the definition of RECIST v1.1.
8. Physical fitness score ECOG 0 or 1 point
9. Toxicity of previous antitumor therapy has returned to ≤ level 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic laboratory abnormalities considered by the investigators, such as elevated ALP, hyperuricemia, and elevated blood glucose; Toxicities with no safety risk, such as hair loss and grade 2 peripheral neurotoxicity, were excluded. Or decreased hemoglobin except ≥90 g/L).
10. No serious cardiac dysfunction, left ventricular ejection fraction (LVEF) ≥50%
11. The organ function level must meet the following requirements: a) bone marrow function: absolute neutrophilic granulocyte count (ANC) ≥1.5×109/L, platelet count ≥90×109/L, hemoglobin ≥90 g/L; b) Liver function: total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN in patients without liver metastasis, AST and ALT ≤5.0 ULN in patients with liver metastasis; c) Kidney function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula).
12. Coagulation function: International normalized ratio (INR)≤1.5×ULN, and activated partial thromboplastin time (APTT)≤1.5ULN.
13. Urinary protein ≤2+ or ≤1000mg/24h.
14. For premenopausal women with childbearing potential, a pregnancy test must be taken within 7 days prior to the start of treatment. Serum or urine pregnancy must be negative and must be non-lactating; all participants (regardless of male or female) in the group should be treated throughout the treatment. Adequate barrier contraceptive measures should be taken during the treatment and 6 months after the treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, major surgery, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration; oral fluorouracil-like drugs such as S-1, capecitabine, or palliative radiotherapy within 2weeks prior to the first administration.
2. Participants with history of severe heart disease, such as: symptomatic congestive heart failure (CHF) ≥ grade 2 (CTCAE 5.0), New York Heart Association (NYHA) ≥ grade 2 heart failure, history of transmural myocardial infarction, unstable angina pectoris etc.
3. Participants with prolonged QT interval (male QTc> 450 msec or female QTc> 470 msec), complete left bundle branch block, III grade atrioventricular block.
4. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for type I diabetes, hypothyroidism that can be controlled only by alternative treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis).
5. Other malignant tumors were diagnosed within 5 years prior to the first administration with the following exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after radical resection.
6. Participants with poorly controlled hypertension by two kinds of antihypertensive drugs (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg).
7. Participants have grade 3 lung disease defined according to NCI-CTCAE v5.0, or a history of interstitial lung disease (ILD).
8. Unstable thrombotic events such as deep vein thrombosis, arterial thrombosis and pulmonary embolism requiring therapeutic intervention within 6 months prior to screening; Thrombus formation associated with infusion set is excluded.
9. Symptoms of active central nervous system metastasis. However, patients with stable brain parenchymal metastases can be enrolled. Stable was defined as: a. The seizure-free state lasted for > 12 weeks with or without the use of antiepileptic drugs; b. Glucocorticoid use is not required; c. Consecutive MRI scans (at least 8 weeks between scans) showed stable imaging status.
10. Patients with a history of allergy to recombinant humanized antibody or mouse chimeric antibody or to any excipients of BL-B01D1.
11. Previous recipients of organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
12. In previous adjuvant therapy with anthracyclines, the cumulative dose of anthracyclines was > 360 mg/m2.
13. Positive human immunodeficiency virus antibody (HIVAb), active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 103 IU/ml) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower limit of detection).
14. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, septicemia, etc.
15. Participated in another clinical trial (calculated from the time of the last dose) within 4 weeks prior to the first dose.
16. The other conditions of participation in this clinical trial were not considered appropriate by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1 .
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of BL-B01D1 will be investigated.
AUC0-t | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to 21 days after the first dose
  CL in the serum of BL-B01D1 per unit of time will be investigated.
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Incidence and titer of ADA of BL-B01D1 will be evaluated.
Nab (neutralizing antibody) | Up to approximately 24 months
  Incidence and titer of Nab of BL-B01D1 will be evaluated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PHD, Principal Investigator — Sun Yat-sen University
Locations (8):
- China (8):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi

REFERENCES:
- [Derived] Ma Y, Huang Y, Zhao Y, Zhao S, Xue J, Yang Y, Fang W, Guo Y, Han Y, Yang K, Li Y, Yang J, Fu Z, Chen G, Chen L, Zhou N, Zhou T, Zhang Y, Zhou H, Liu Q, Zhu Y, Zhu H, Xiao S, Zhang L, Zhao H. BL-B01D1, a first-in-class EGFR-HER3 bispecific antibody-drug conjugate, in patients with locally advanced or metastatic solid tumours: a first-in-human, open-label, multicentre, phase 1 study. Lancet Oncol. 2024 Jul;25(7):901-911. doi: 10.1016/S1470-2045(24)00159-1. Epub 2024 May 29. PMID 38823410